CLINICAL TRIAL: NCT04699630
Title: A Phase II Study of U3-1402 (Patritumab Deruxtecan) in Patients With Metastatic Breast Cancer
Brief Title: A Study of U3-1402 (Patritumab Deruxtecan) in Subjects With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BRE 354
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer
Keywords: Breast Neoplasm; HER3 Expression; Hormone Receptor Positive Breast Cancer; Triple Negative Breast Cancer; Metastatic breast cancer; locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Participants will receive 5.6 mg/kg U3-1402 (Patritumab Deruxtecan) intravenously on day 1 every 3 weeks. All participants will undergo pre-treatment biopsies. (An archival tissue sample taken within two months of treatment should be provided if it is not medically feasible to provide a pre-treatment biopsy). Up to 60 participants will be enrolled into this arm.
  Interventions: Drug: U3-1402
- Part B (Experimental): Participants will receive 5.6 mg/kg U3-1402 intravenously on day 1 every 3 weeks. Part B will enroll 20 participants with metastatic hormone-receptor positive (HR+) HER2-negative cancer and 20 participants with metastatic triple-negative breast cancer (mTNBC), regardless of HER3 expression.
  Interventions: Drug: U3-1402
- Part Z (Experimental): Participants will receive 5.6 mg/kg U3-1402 (Patritumab Deruxtecan) intravenously on day 1 every 3 weeks. Part Z will enroll an additional 21 participants with HER2+ MBC.
  Interventions: Drug: U3-1402

INTERVENTIONS:
Drug: U3-1402 — All subjects will receive 5.6 mg/kg U3-1402 (Patritumab Deruxtecan) intravenously on day 1 of every 3 weeks. One cycle is defined as 3 weeks.
  Other Names: Patritumab Deruxtecan

SUMMARY:
This study is to evaluate safety and efficacy of an antibody drug conjugate U3-1402 (patritumab deruxtecan) in patients with locally advanced or metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
U3-1402 (Patritumab Deruxtecan) is an antibody drug conjugate comprising a recombinant fully human anti HER3 monoclonal antibody linked to a linker containing topoisomerase I inhibitor. This is a phase II study of U3-1402 (patritumab deruxtecan) in subjects with MBC. The study will be conducted in 3 parts (Part A , Part B, and Part Z). All enrolled subjects in Part A will undergo pretreatment biopsies to determine if subjects with particular biomarker expression (ER/PR/HER2/HER3) show preliminary efficacy. Part B will enroll subgroups of participants that are metastatic, hormone receptor-positive (HR+) HER2-negative or triple-negative (mTNBC) regardless of HER3 expression that were defined from Part A analysis. Part Z will enroll participants with HER2- positive (HER2+) MBC.

ELIGIBILITY:
Eligibility Criteria:

Inclusion criteria for Part A and B (HER2-negative) and Part Z (HER2-positive) cohorts:

1. Written informed consent, according to local guidelines, signed and dated by the patient or by a legal guardian prior to the performance of any study-specific procedures, sampling, or analyses
2. Women and men at least 18 years-of-age at the time of signature of the informed consent form (ICF)
3. Histologically documented locally advanced or metastatic breast cancer
4. Triple-negative breast cancer (TNBC) patients should have received at least 1 but no more than 5 prior lines of chemotherapy in the metastatic setting
5. Parts A and B patients only: Patients with HR+ HER2-negative MBC should have received prior treatment with endocrine therapy +CDK 4/6 inhibitor. No limit to prior endocrine therapy regimens, but no more than 2 prior chemotherapy regimens in the metastatic setting are allowed. HR+ = Estrogen receptor (ER) and/or Progesterone (PgR) positivity that are defined as ≥1% of cells expressing HR via IHC analysis. HER2 negativity is defined as either of the following: IHC 0, IHC 1+, or IHC 2+/in situ hybridization (ISH) negative.
6. Part B patients only: Patients with HER2-negative MBC will be included into one of the following 2 subgroups: 1) MBC HR+, HER2-, regardless of HER3 expression, who have received trastuzumab deruxtecan and/or sacituzumab govitecan, or, 2) mTNBC, regardless of HER3 expression, who have received sacituzumab govitecan and/or datopotamab deruxtecan.
7. Part Z patients only: should have documented HER2-positive expression as per American Society of Clinical Oncology - College of American Pathologists guidelines based on local testing.
8. Part Z patients only: should have had prior treatment with at least 2 anti-HER2 therapies, 1 of which must be trastuzumab deruxtecan. These patients must have experienced disease progression after receiving trastuzumab deruxtecan.
9. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (bone-only disease excluded)
10. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed ≥4 weeks prior to initiation of study treatment (2 weeks for patients who received palliative radiation therapy), there is no evidence of central nervous system disease progression on a scan or mild neurologic symptoms, and there is no requirement for chronic corticosteroid therapy for the treatment of brain metastases
11. Willingness to undergo pre-treatment biopsy and on-treatment biopsies; must have a tumor amenable to pre-treatment biopsy (unless archived tissue is available and was obtained within 2 months prior to starting treatment) and on-treatment biopsy (excludes bone lesions and previously irradiated lesions)
12. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
13. Has adequate organ function within 7 days before the start of study treatment, defined as:

    * Platelet count ≥100 × 109/L
    * Hemoglobin (Hb) ≥9 g/dL (transfusion and/or growth factor support allowed)
    * Absolute neutrophil count ≥1.5 × 109/L
    * Prothrombin time (PT) and partial thromboplastin time (PTT) ≤1.5 × the upper limit of normal (ULN), except for patients on coumadin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-international normalized ratio (INR) within therapeutic range as deemed appropriate by the Investigator
    * Serum creatinine ≤1.5 × ULN, or creatinine clearance ≥50 mL/min as calculated using the modified Cockcroft-Gault equation; confirmation of creatinine clearance is only required when creatinine is >1.5 × ULN
    * AST/ALT ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
    * Total bilirubin ≤1.5 × ULN if no liver metastases or <3 × ULN in the presence of documented Gilbert's syndrome or liver metastases
    * Serum albumin ≥2.5 g/dL
14. Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for at least 7 months following last dose. Male patients must also refrain from donating sperm during their participation in the study.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from study entry:

Exclusion criteria for Parts A and B (HER2-negative) and Part Z (HER2-positive) cohorts:

1. Treatment with any of the following:

   * Any systemic anti-cancer chemotherapy, small molecule, biologic, hormonal agent, or immune checkpoint inhibitor therapy from a previous treatment regimen or clinical study within 21 days prior to the first dose of patritumab deruxtecan
   * Prior treatment with any HER3-targeting agent
   * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug treatment
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug treatment, or palliative radiation therapy within 2 weeks of the first dose of study drug treatment
   * Chloroquine /hydroxychloroquine ≤14 days prior to the first dose of study drug treatment
2. Has any hypersensitivity to drug substances or inactive ingredients in drug product
3. Has any history of ILD (including pulmonary fibrosis or radiation pneumonitis), has clinically significant ILD, or is suspected to have such disease by imaging during screening. If imaging findings are unlikely to indicate a history of pneumonitis, then the Investigator should discuss the considerations with the Medical Monitor about potential enrollment and record the reasoning in the source documentation.
4. Clinically severe pulmonary compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

   * Any underlying pulmonary disorder (e.g., pulmonary emboli, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion)
   * Any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis)

   OR prior pneumonectomy
5. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or baseline at the time of starting study treatment. Note: patients with chronic Grade 2 toxicities who are asymptomatic or adequately managed with stable medication may be eligible with approval by the Medical Monitor.
6. Leptomeningeal metastases or evidence of spinal cord compression or brain metastases, defined as being clinically active and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Patients with clinically inactive or treated brain metastases who are asymptomatic (i.e., without neurologic signs or symptoms and do not require treatment with corticosteroids or anticonvulsants) may be included in the study. Patients must have a stable neurologic status for at least 2 weeks prior to Cycle 1 Day 1.
7. Women who are pregnant, nursing, or plan to become pregnant while in the study and for at least 7 months after the last administration of study treatment
8. Men who plan to father a child while in the study and for at least 7 months after the last administration of study treatment
9. Uncontrolled or significant cardiovascular disorder prior to Cycle 1 Day 1, including:

   * Mean resting corrected QT interval using Fridericia's formula (QTcF) prolongation to >470 ms for females and >450 ms for males in three successive screening measurements
   * Patients with a left ventricular ejection fraction (LVEF) <50%
   * Resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).
   * Documented myocardial infarction within 6 months
   * Congestive heart failure (New York Heart Association ≥ Grade 2 within 28 days
10. Has known clinically significant corneal disease from prior therapies such as drug-induced keratitis
11. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Patients who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
12. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection, including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
13. Presence of other active invasive cancers other than the one treated in this study within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment
14. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol

    Additional exclusion criteria only for Parts A and B (HER2-negative) cohorts:
15. Patients with HER2+ breast cancer per ASCO-CAP guidelines
16. Part A only: Prior treatment with an antibody drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g., trastuzumab deruxtecan, DS-1062a [datopotamab deruxtecan], and DS-7300a [B7-H3 DXd-ADC])
17. Part B patients only: Prior treatment with trastuzumab deruxtecan, sacituzumab govitecan, and/or datopotamab deruxtecan with any of the following:

    * A severe reaction or severe tolerability issues that necessitated stopping treatment with the therapy
    * Any unresolved toxicities from the prior therapy greater than Grade 1, with the exception of alopecia

    Additional exclusion criteria only for Part Z (HER2-positive) cohort:
18. Treatment with any of the following:

    * Prior treatment with an antibody drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor except trastuzumab deruxtecan
    * Prior treatment with trastuzumab deruxtecan within 4 weeks prior to the first dose of patritumab deruxtecan
19. Uncontrolled or significant cardiovascular disease, including history of myocardial infarction within 6 months before enrollment
20. A severe reaction or severe tolerability issues that necessitated stopping treatment with trastuzumab deruxtecan
21. Any unresolved toxicities from prior therapy with trastuzumab deruxtecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) of single agent U3-1402 (patritumab deruxtecan) in participants with MBC | Assessed every 6 weeks for the first 6 months then every 9 weeks thereafter until disease progression or death or up to 33 months.
  ORR is defined as the proportion of participants with confirmed complete response (CR) or partial response (PR) (i.e., confirmation at least 4 weeks apart) according to RECIST Version 1.1 criteria.
  Per RECIST V1.1: A CR is defined as disappearance of all target and non-target lesions. A PR is defined as ≥30% decrease in the sum of diameters of target lesions from baseline sum.
Rate of participants without disease progression at 6 month to determine six-months Progression Free survival (PFS-6) of single agent U3-1402 (patritumab deruxtecan) in participants with MBC | Every 6 weeks after day 1 for the first 6 months
  PFS-6 is defined as the rate of participants without disease progression (PD) at six months from the start of study drug according to RECIST version 1.1 criteria.
  Per RECIST V1.1, a PD is ≥20% increase in target lesions and ≥5mm from smallest sum, appearance of any new lesions, or unequivocal progression of non-target lesions

SECONDARY OUTCOMES:
Incidence of participants with adverse events to assess the safety and tolerability of U3-1402 (patritumab deruxtecan) in participants with MBC | From day 1 until 40 days after end of treatment or up to 33 months
  Safety is determined by proportion of participants who experience adverse events and serious adverse events when given U3-1402.
Median Duration of Response (DOR) in participants with MBC | Assessed every 6 weeks for the first 6 months then every 9 weeks thereafter until disease progression or death or up to 33 months.
  Duration of response (DOR) is defined as the duration from the first documented response to the date of disease progression (PD) according to the RECIST V1.1 criteria or death due to any cause.
  Per RECIST V1.1, a PD is ≥20% increase in target lesions and ≥5mm from smallest sum, appearance of any new lesions, or unequivocal progression of non-target lesions
Median Progression-Free Survival (PFS) in participants with MBC | Assessed every 6 weeks for the first 6 months then every 9 weeks thereafter until disease progression or death or up to 33 months
  Progression Free Survival (PFS) is defined as the time from start of study treatment to the date of the first documented disease progression (PD) according to the RECIST V1.1 criteria or death due to any cause.
  Per RECIST V1.1, a PD is ≥20% increase in target lesions and ≥5mm from smallest sum, appearance of any new lesions, or unequivocal progression of non-target lesions
Clinical Benefit Rate (CBR) in participants with MBC | Assessed every 6 weeks for the first 6 months then every 9 weeks thereafter until disease progression or death or up to 33 months
  CBR is defined as the rate of participants with CR, PR, or best overall response of SD for ≥ 6 months according to the RECIST v 1.1 criteria Per RECIST V1.1: A CR is defined as the disappearance of all target and non-target lesions. A PR is defined as ≥30% decrease in the sum of diameters of target lesions from the baseline sum. An SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Overall response rate (ORR) of single agent U3-1402 (patritumab deruxtecan) in participants with HER2+ MBC after progression on trastuzumab deruxtecan | Assessed every 6 weeks for the first 6 months then every 9 weeks thereafter until disease progression or death or up to 33 months
  ORR is defined as the rate of participants with confirmed complete response (CR) or partial response (PR) (i.e., confirmation at least 4 weeks apart) according to RECIST Version 1.1 criteria.
  Per RECIST V1.1: A CR is defined as disappearance of all target and non-target lesions. A PR is defined as ≥30% decrease in the sum of diameters of target lesions from baseline sum.
Rate of participants without disease progression at 6 month to determine six-months Progression Free survival (PFS-6) of single agent U3-1402 (patritumab deruxtecan) in participants with HER2+ MBC after progression on trastuzumab deruxtecan | Every 6 weeks after day 1 for the first 6 months
  PFS-6 is defined as the rate of participants without disease progression (PD) at six months from the start of study drug according to RECIST version 1.1 criteria.
  Per RECIST V1.1, a PD is ≥20% increase in target lesions and ≥5mm from smallest sum, appearance of any new lesions, or unequivocal progression of non-target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hamilton, MD, Study Chair — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Highlands Oncology Group, Springdale, Arkansas
  - City of Hope, Duarte, California
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers-Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No